CLINICAL TRIAL: NCT00983749
Title: A Randomized, Controlled Phase 1 Study of External Counterpulsation as a Treatment for Acute Ischemic Stroke
Brief Title: Safety Study of External Counterpulsation as a Treatment for Acute Ischemic Stroke
Acronym: CUFFS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Alabama at Birmingham (Other); University of California, Los Angeles (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Kama Guluma, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPOTRIAS Project 1; 3P50NS044148-06S1 (NIH)
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Stroke
Keywords: External Counterpulsation; Counterpulsation, Diastolic; Ultrasonography, Doppler, Transcranial; Blood Flow Velocity; Neurologic Deficit
MeSH Terms: conditions — Stroke; Heart Murmurs; Neurologic Manifestations | interventions — Counterpulsation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full-pressure ECP (Experimental): Patients in the "Full-pressure ECP" arm receive a 1-hour treatment of ECP at full pressure, which will be applied in a tiered, dose-escalating manner up to 300mmHg, while assessments are made.
  Interventions: Device: Full-pressure ECP
- Sham-pressure ECP (Sham Comparator): A 1-hour treatment of ECP at an inactive pressure (75mmHg)
  Interventions: Device: Sham-pressure ECP

INTERVENTIONS:
Device: Full-pressure ECP — A one-hour treatment of ECP at full pressure, which will be applied in a tiered, dose-escalating manner, starting at 200mmHg and increasing up to 300mmHg based on assessments made.
  Other Names: External counterpulsation
  Arms: Full-pressure ECP
Device: Sham-pressure ECP — A one-hour treatment of ECP at an inactive pressure, which will be applied at 75mmHg and kept there for the hour while assessments are made.
  Other Names: External counterpulsation
  Arms: Sham-pressure ECP

SUMMARY:
The purpose of this study is to determine if external counterpulsation (ECP) is feasible to perform, tolerable, and safe as a treatment for patients with acute ischemic stroke (i.e., a blockage of one of the arteries supplying a part of the brain), and to assess what type of effect it might have on 1) the velocity of blood flow in the arteries supplying the brain and 2) stroke symptoms. The hypothesis of the study is that ECP will be feasible and safe to perform, and will be tolerable for patients with acute ischemic stroke at pressures that increase the velocity of arterial blood flow to the brain.

DETAILED DESCRIPTION:
A stroke is usually caused by a blockage of one of the arteries that carries blood to the brain. Sometimes with a stroke, there may be a small amount of blood flow that manages to get through or around the blockage, and it may be possible that the amount of damage from a stroke may be reduced by increasing this blood flow. External counterpulsation (ECP) is a procedure in which a machine uses electrical signals from the heart that are detectable on the surface of the body in order to time the inflation of cuffs (similar to a blood pressure cuff) that are wrapped around a patient's legs (calves, thighs and buttocks). Using a reading of the electrical activity from the patient's heart (an electrocardiogram, or ECG, monitor), the machine inflates the cuffs with air at just the right time during each heart beat, during diastole, in order to change the blood pressure in a way that has been shown to increase blood flow to the kidneys, skin, eyes, heart, and brain.

In this study, patients presenting within the first 48 hours of an acute ischemic stroke (i.e., a blockage of one of the arteries supplying a part of the brain) will be randomly assigned to either of (1) a 1-hour treatment of external counterpulsation (ECP) applied at a pressure that is typically therapeutic, or (2) a 1-hour treatment of ECP at a minimal pressure in a control group. ECP-induced changes in brain artery flow velocity will be assessed with an ultrasound prior to and then during ECP in each group, and an optimal pressure that results in an augmentation of flow velocity will be determined. A neurological exam will be performed prior to, during, and after ECP in each group, in order to assess any changes in stroke symptoms related to ECP. Patients will be followed to 30 days. The main goal of this trial is to evaluate if ECP is safe and feasible to use as a treatment for stroke. In addition, the trial will enable an assessment of whether or not ECP increases blood flow to the brain or affects the neurological symptoms of a patient with a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 85, inclusive
* Symptoms consistent with acute ischemic stroke, with a measurable neurological deficit at presentation
* Ability to initiate external counterpulsation within 48 hours of stroke onset
* No evidence of hemorrhage on CT scan or MRI
* MCA distribution stroke: a total or partial anterior circulation infarct (TACI or PACI by Oxfordshire criteria) consistent with MCA distribution ischemia, or a lacunar stroke felt by the investigator to possibly involve a deep perforating branch in the MCA territory (LACI by Oxfordshire criteria)

Exclusion Criteria:

* Rapidly resolving stroke symptoms consistent with a transient ischemic attack
* Severe stroke defined as an NIHSS > 22
* Intracranial hemorrhage (SAH, EDH, SDH, IPH, hemorrhagic conversion) on CT scan
* Brain tumor or brain abscess on CT scan or MRI
* Presentation consistent with subarachnoid hemorrhage (such as a sudden, severe thunderclap headache, or an associated third nerve palsy)
* History of cerebral aneurysm, AVM, or hemorrhagic stroke
* Either treatment or planned treatment of current stroke with standard thrombolytic therapy (intravenous or intra-arterial) or neurothrombectomy
* History of lower limb amputation above the ankle
* History of untreated aortic dissection
* History or suspicion of thoracic or abdominal aortic aneurysm
* Known significant anomaly of the heart, aorta, or great vessels that would be complicated by elevated diastolic pressures.
* BP > 180/100 that remains so after minimal treatment (such as one or two doses of an antihypertensive agent, or as determined by the investigator)
* History of non-trivial aortic regurgitation, or any symptomatic valvular heart disease determined by the investigator to be at risk of worsening on ECP
* Significant symptomatic congestive heart failure (orthopnea, CHF-related dyspnea, or rales and jugular venous distention on exam) or a left ventricular ejection fraction known to be <30%
* Diagnosis of significant lower extremity peripheral vascular occlusive disease (PVOD), or symptomatic PVOD as determined by the investigator (especially symptoms of claudication)
* Phlebitis, stasis ulcer, severe varicosities
* Diagnosis of DVT within the past month, or current symptoms strongly suggestive of new DVT, such as asymmetric calf or leg swelling, discomfort, or erythema (to be evaluated by screening duplex)
* Pacemaker or automated implanted defibrillator (AICD)
* A cardiac dysrhythmia (such as atrial fibrillation or atrial flutter, or frequent premature ventricular contractions (PVCs) or premature atrial contractions (PACs) as determined by the investigator) that would interfere with ECP triggering
* Pregnancy (as determined by a urine pregnancy test in females of child-bearing age)
* Known coagulopathy, thrombocytopenia with platelet count < 100,000, or taking warfarin with an INR > 2.0.
* History positive for chronic low back pain, radiculopathy suggestive of herniated lumbar disc, or related surgery
* Known collagen vascular disease
* Obesity to a degree (as determined by the investigator) that would prevent proper placement and/or activation of counterpulsation cuffs
* Any psychological, social, or legal condition that would interfere with the ability of the patient or his or her surrogate to give Informed Consent and/or his or her capacity to comply with all study requirements, including the necessary time commitment
* An inadequate temporal window for TCD insonation.
* Currently involved or have been involved in a clinical trial within the last 30 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-12; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kama Z Guluma, M.D., Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - University of Alabama Hospital, Birmingham, Alabama
  - UCLA Medical Center, Los Angeles, California
  - UCSD Medical Center, San Diego, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 23 patients with symptoms and signs of acute middle cerebral artery (MCA) ischemic stroke presenting within 48 hours of onset at three academic medical centers in the United States.
Pre-assignment Details: Before randomization, all patients underwent duplex ultrasound scanning of the legs to rule out deep vein thrombosis (DVT), along with an assessment of temporal window adequacy for transcranial doppler (TCD); patients meeting these criteria were randomly assigned to one of two treatment arms (all the patients that were enrolled met these criteria).
Groups:
- Full-pressure ECP: Patients in the "Full-pressure ECP" arm received a 1-hour treatment of ECP at full pressure, applied in a tiered, dose-escalating manner up to 300mmHg, while assessments were made.
- Sham-pressure ECP: Patients receiving sham-pressure ECP received a one-hour treatment of ECP at an inactive pressure, applied at 75mmHg and kept there for the hour while assessments were made.
Period: Acute Phase (Enrollment to Hospital DC)
Arm/Group | Full-pressure ECP | Sham-pressure ECP
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0
Period: Follow-up Phase (Hospital DC to 30 Days)
Arm/Group | Full-pressure ECP | Sham-pressure ECP
Started | 13 | 10
Completed | 12 | 7
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full-pressure ECP | Sham-pressure ECP | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [50 to 66] | 57 [55 to 60] | 57 [52 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Tolerability of External Counterpulsation
Description: The first primary outcome measure was tolerability and feasibility. Tolerance was defined as the absence of any indications to stop the procedure or reduce the pressure to a non-therapeutic level. Feasibility was defined in the full-pressure group as the sustained (at least 30 minutes) tolerance of any pressure capable of causing a 15% augmentation of MFV in 90% of subjects, and defined in the sham-pressure group as the sustained tolerance of the sham pressure in all subjects.
Time Frame: During one hour of treatment
Measure: Number; unit: participants
Arm/Group | Full-pressure ECP | Sham-pressure ECP
Number analyzed (Participants) | 13 | 10
participants | 12 | 9

2. Primary Outcome: Safety (Including Endpoints Such an Increase NIHSS During or Immediately After ECP, and Acute Hemorrhage on Repeating Imaging, Serious Adverse Events Related to ECP, Mortality)
Description: Safety was evaluated by the incidence of serious adverse events (SAEs) or acute neurological deterioration in relation to the study device and/or procedures at 30 days, the incidence of acute symptomatic hemorrhage on repeat imaging at 24 hours, the incidence of all adverse events (AEs) in the first 48 hours, and mortality at 30 days. The National Institutes of Health Stroke Scale (NIHSS) is a stroke severity scale, based on examination, that goes from 0 (no deficit) to a maximum of 42. Acute neurological deterioration - which was captured as a serious adverse event - was defined as a ≥4-point increase on the NIHSS, or a ≥2-point decline in level of consciousness item 1a on the NIHSS, or a new neurological deficit, or clinically significant worsening of motor function lasting more than 8 hours and attributable to a neurological entity. Symptomatic intracranial hemorrhage was defined as new hemorrhage on CT that was associated with acute neurological deterioration.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Full-pressure ECP | Sham-pressure ECP
Number analyzed (Participants) | 13 | 10
participants
  Patients with at least one AE | 12 | 8
  Patients with device or treatment-related SAE | 0 | 0
  Symptomatic hemorrhage at 24 hour | 0 | 0
  Acute neurological deterioration | 0 | 0
  Deaths reported out to 30 days | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected out to 48 hours, and Serious Adverse Events (SAEs) were collect out to 30 days.
Arm/Group | Full-pressure ECP | Sham-pressure ECP
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/10
Other Adverse Events (participants affected / at risk) | 12/13 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full-pressure ECP (N=13) | Sham-pressure ECP (N=10)
Transient ischaemic attack (Nervous system disorders) | 1 (2) | 0 (0)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full-pressure ECP (N=13) | Sham-pressure ECP (N=10)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Carotid artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No